CLINICAL TRIAL: NCT05832580
Title: The Prevention of Systemic Ectopic Mineralization in Pseudoxanthoma Elasticum
Acronym: TEMP-PREVENT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Wilko Spiering, MD, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-552
Record Dates: First submitted 2023-03-14; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Pseudoxanthoma Elasticum
MeSH Terms: conditions — Pseudoxanthoma Elasticum | interventions — Etidronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etidronate (Experimental): Daily dosis of 20mg/kg of etidronate in a cyclical regimen of 2 weeks on and 10 weeks off, for a total of 24 months.
  Interventions: Drug: Etidronate
- Placebo (Placebo Comparator): Daily dosis of placebo in a cyclical regimen of 2 weeks on and 10 weeks off, for a total of 24 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etidronate — Etidronate in capsules of 200 mg or 400 mg.
  Arms: Etidronate
Drug: Placebo — Placebo in similar capsules
  Arms: Placebo

SUMMARY:
The goal of this randomized clinical trial is to assess the effect of etidronate on ectopic calcification in relatively young patients with Pseudoxanthoma elasticum. The main question it aims to answer are:

What is the difference in the arterial calcification scores in the legs and the carotid syphon measured on low-dose CT scan after 24 months of treatment compared to baseline between etidronate and placebo.

Participants will be asked to do take etidronate or placebo for 24 months.

DETAILED DESCRIPTION:
SUMMARY Rationale: Pseudoxanthoma elasticum is a monogenic disease caused by mutations in the ABCC6 gene. These mutations result in reduced levels of inorganic pyrophosphate, a strong inhibitor of ectopic calcification. This loss of inorganic pyrophosphate leads to a typical pattern of progressive degradation and calcification of elastin fibers in the skin, the medial layer of small- and medium sized arteries and the Bruch's membrane of the retina. This results clinically in skin disorders (pseudoxanthoma's), peripheral arterial disease, gastric bleeding and stroke. The progressive calcification of the Bruch's membrane in the retina results in peau d' orange, angioid streaks, choroidal neovascularizations (CNV's) and macular atrophy. Due to this eye pathology, PXE results in visual impairment and legal blindness at a young age.

The bisphosphonate etidronate is a molecular homologue of pyrophosphate, which therefore has the potential to substitute the loss of pyrophosphate that is seen in PXE. It has been on the market for over 40 years and has a well-established safety profile. Based upon positive results from animal studies, studies in related genetic disorders, and trials in patients with renal disease, recently a double blind, randomized, placebo-controlled clinical trial (RCT) in PXE patients was conducted. This Treatment of Ectopic Mineralization in PXE (TEMP)-trial (protocol ID: NL47602.041.15) showed that one year of treatment with etidronate was safe, and reduced calcifications of the leg arteries and of other vascular beds compared to placebo in PXE patients with arterial calcifications. As no other systemic treatment for PXE exists, this established etidronate as a very promising therapeutic option. The TEMP trial focused on reduction of complications in symptomatic patients with arterial calcifications (mean age 57). Since arterial calcification are so common in PXE patients, the vascular diseases associated with them are as well much more prevalent in the PXE population compared to the general population.

The aim of the TEMP-PREVENT is to include younger patients who developed no or only little vascular calcifications. The investigators suspect that the formation of calcium deposits can be halted in the intima for a large part, if not all together. If so, PXE patients would have the same vascular risk profiles as their peers.

Objective: Primary aim:

To investigate the effect of etidronate on arterial calcification, and therefore vascular health.

Secondary aims:

To investigate the effect of etidronate on ophthalmological measures (including calcifications in Bruch's membrane), dermatological measurements, laboratory measurements, vascular measurements, incidence of major adverse cardiovascular events (MACEs), safety measures, and quality of life.

Study design: Double blind, placebo controlled, randomized clinical trial

Study population: Patients with a confirmed diagnosis of pseudoxanthoma elasticum from 18 - 50 years old.

Intervention: One group receives daily a dosis of 20mg/kg of etidronate in a cyclical regimen of 2 weeks on and 10 weeks off, for a total of 24 months. The other group receives a matching placebo with the same cyclical regimen and duration.

Main study endpoints: Primary endpoint:

The mean difference in the arterial calcification scores in the legs and the carotid syphon measured on low-dose CT scan after 24 months of treatment compared to baseline between etidronate and placebo.

Secondary endpoints:

Differences in Bruch's membrane reflectivity on high-definition spectral domain optical coherence tomography (HD-OCT); OCT-angiography; ophthalmological measures (visual acuity, fundus photography and autofluorescence), dermatological measurements (elastin degradation and calcification), measurement of pyrophosphate and desmosine, vascular measurements (calcification on CT, carotid intima thickness (cIMT), pulse wave velocity (PWV), ankle brachial index (ABI), WELCH questionnaire and the six-minute walking test), intracranial pulsatility and vascular anatomy on MRI, incidence of MACEs, quality of life (EQ-5D), and safety measures (calcium, phosphate, number of anti-VEGF injections), after 24 months of treatment compared to baseline between etidronate and placebo.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Each patient will visit the University Medical Center Utrecht (UMCU) four times during the study (screening, M0, M12, M24). A low dose scan of the head and the legs (M0, M24) will be made, for which the effective dosage of radiation is approximately 1.42 mSv in for a person with a weight of 70kg. The total radiation dosage for the study is therefore, approximately, 2.84 mSv. Theoretically, this radiation dose could increase the risk of future cancer. For ophthalmological assessments (M0, M12, M24), standard ophthalmological examination in combination with an OCT scan, will be performed, which yield no additional harm apart from the mydriatic eye drops. Dermatological assessments will be carried out by a punch biopsy of the skin (M0, M24), and laboratory assessments by venepuncture (M0, M12, M24), which, besides the normal risk associated with these procedures (hematoma, tenderness and swelling, persistent bleeding, vasovagal response, infection, hypersensitivity for anaesthesia) yield no additional harm. Given the well-established safety profile of etidronate and our experience from the TEMP trial, the investigators deem the overall risk of this trial to be low. The aim of this trial is to investigate the preventive effects of etidronate in PXE patients early in the disease. Given that we currently treat patients with etidronate only when arterial calcifications have already manifested, there is a potential clinical benefit to be gained by participation in this trial. Given the inhibitory effect of etidronate on arterial calcifications, it is expected that the TEMP-PREVENT trial opens new treatment possibilities for younger PXE patients.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* 1. Be between 18 years and 50 years.
* 2. Have a definitive diagnosis of PXE according to the Plomp criteria, which confirm a diagnosis of PXE when at least two (or more) criteria not belonging to the same category (skin, eye, genetic) are met:

  1. Skin

     1. Yellowish papules and/or plaques on the lateral side of the neck and/or flexural areas of the body or
     2. Increase of morphologically altered elastin with fragmentation, clumping and calcification of elastic fibers in a skin biopsy taken.
  2. Eye

     1. Peau d'orange of the retina or
     2. One or more angioid streaks (AS), each at least as long as one disk diameter. When in doubt, fluorescein or indocyanine green angiography of the fundus is needed for confirmation.
  3. Genetics

     1. A pathogenic mutation of both alleles of the ABCC6 gene or
     2. A first-degree relative (parent, sibling or child) who meets independently the diagnostic criteria for definitive PXE
* 3. Fertile women must take adequate anticonception.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Patients that are unable or unwilling to sign for informed consent.
2. Pregnant, lactating, or fertile women who might wish to become pregnant within three years.**
3. Patients with an estimated glomerular filtration rate below 30 ml/min/1.73m2 according to the CKD-EPI equation.31
4. Patients with a known abnormality of the oesophagus that would interfere with passage of the drug (e.g. oesophagus stenosis).
5. Patients with chronic diarrhoea (> 1 month).
6. Patients with known osteomalacia;
7. Patients with hypocalcaemia (calcium <2.20 mmol/L corrected for albumin)*.
8. Patients with a vitamin D deficiency (<35 nmol/L)*.
9. Patients that used a bisphosphonate in the last 5 years.
10. Patients with known sensitivity to etidronate.
11. Any other medical or social condition that, at the discretion of the Principal Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data.

    * After correction a patient is again suitable for participation, as long as inclusion criteria are met (more information in paragraph 7.3.3).

      * Subjects that become pregnant during the trial will be excluded from further participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-04-26 (Estimated); Primary Completion 2027-03-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Arterial calcification | 24 months.
  The difference in arterial calcification volume measured (uL) on CT-scans between the etidronate and placebo group 24 months.

SECONDARY OUTCOMES:
Ophtalmology: Visual acuity | 24 months.
  Difference in visual acuity at phtalmologic exam.
Ophtalmology: Contrast sensitivity. | 24 months.
  Difference in contrast sensitivity at ophtalmologic exam.
Ophtalmology: Reflectivity of Bruch's membrane | 24 months.
  Difference in normalized reflectivity in Bruch's membrane as measured with SD-optical coherence tomography, between the etidronate and placebo group after 24 months.
Ophtalmology: Length of angioid streaks. | 24 months.
  Length of angioid streaks in the fundus, between the etidronate and placebogroup after 24 months.
Ophtalmology: Area of angioid streaks. | 24 months.
  Amount of area coverd by angioid streaks in the fundus, between the etidronate and placebogroup after 24 months.
Ophtalmology: Area of atrophy | 24 months.
  The area of artophy on near-Infrared between etidronate an de placebogroup after 24 months.
Intra cranial velocity pulsatility index on MRI | 24 months.
  Difference in the intracranial velocity pulsatility index as measured with MRI, between the etidronate and placebo group after 24 months.
Elastin degradation of the skin | 24 months.
  Difference in the amount of elastin degradation in the skin in observation of skin biopsies, between the etidronate and placebo group after 24 months.
Calcification of the skin | 24 months.
  Difference in the amount of calcified tissue in the skin in observation of skin biopsies, between the etidronate and placebo group after 24 months.
inorganic pyrophosphate | 24 months.
  Difference in plasma inorganic pyrophosphate between the etidronate and placebo group after 24 months.
serum desmosine | 24 months.
  Difference in serum desmosine, between the etidronate and placebo group after 24 months.
Incidence of MACE | 24 months.
  Difference in occurence of major adverse cardiovascular events (stroke, TIA, myocardial infarction or cardiovascular death) between the etidronate and placebo group after 24 months.
EQ-5D | 24 months.
  Difference in reported quality of life, as measured with the EQ-5D, between the etidronate and placebo group after 24 months.
Cognitive Function 15 Words test | 24 months.
  Difference in scores 15 words test between the etidronate and placebo group after 24 months.
Cognitive Function STROOP | 24 months.
  Difference in scores on the STROOP test between the etidronate and placebo group after 24 months.
Cognitive functioning Trailmaking test | 24 months.
  Difference in scores on trailmaking test between the etidronate and placebo group after 24 months.
Cognitive functioning Brixton test | 24 months.
  Difference in scores on brixton test between the etidronate and placebo group after 24 months.
Cognitive Function semantic fluency | 24 months.
  Difference in number of words named in the sematic fluency test between the etidronate and placebo group after 24 months.
Safety: Anti VGEF use | 24 months.
  Difference in number of anti-VEGF injections used, between the etidronate and placebo group after 24 months.
Safety: Plasma calcium | 24 months.
  Difference in plasma calcium (mmol/L) between the etidronate and placebo group after 24 months.
Safety: plasma phosphate | 24 months.
  Difference in plasma phosphate (mmol/L) measured via laboratory assessment, between the etidronate and placebo group after 24 months.
PROMIS 10 | 24 months
  Difference in reported scores on the PROMIS 10 scale between etidronate and placebo after 24 months
PROMIS Physical Funtioning short form | 24 months
  Difference in reported scores on the PROMIS PF scale between etidronate and placebo after 24 months
Utrecht Scale for Evaluation of Rehabilitation | 24 months
  Difference in reported scores on the USER P scale between etidronate and placebo after 24 months
WELCH questionnaire | 24 months
  Difference in reported scores on the WELCH questionnaire between etidronate and placebo after 24 months
6 minute walking test | 24 months.
  Difference distance coverd by walking during the six minute walking test between etidronate and placebo,
Ankle Brachial index | 24 months
  Difference in Ankle Brachial index between etidronate and placebo
Pulse wave velocity (m/s) | 24 months.
  Difference in pulse wave velocity (m/s) between etidronate and placebo.
carotid intima media thickness | 24 months.
  Difference in carotid intima media thickness (um) between etidronate and placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harmsen IM, Haverkamp M, van den Beukel TC, Kok M, de Jong PA, van Valen E, van Leeuwen R, Norel JO, Spiering W. The TEMP-PREVENT trial: a study protocol for a randomized, double-blind, placebo-controlled clinical trial of etidronate for treatment in young adult patients with pseudoxanthoma elasticum. Trials. 2025 Oct 23;26(1):431. doi: 10.1186/s13063-025-09064-6. PMID 41131563